CLINICAL TRIAL: NCT02036853
Title: An Open-Label Trial of Triheptanoin in Patients With Glucose Transporter Type-1 Deficiency Syndrome (GLUT1 DS)
Brief Title: An Open-Label Trial of Triheptanoin in Patients With Glucose Transporter Type-1 Deficiency Syndrome
Acronym: GLUT1DS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adrian Lacy (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Adrian Lacy, Principal Investigator, Cook Children's Health Care System
Organization: Cook Children's Health Care System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-NEUR-001
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Glucose Transporter Type-1 Deficiency Syndrome (Glut1 DS)
Keywords: Triheptanoin; Glut1 DS; Epilepsy; Seizures
MeSH Terms: conditions — Glut1 Deficiency Syndrome; Epilepsy; Seizures | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schedule A (Experimental): Subjects previously treated with triheptanoin
  Interventions: Drug: Triheptanoin
- Schedule B (Experimental): Naïve to triheptanoin
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — Schedule A: Subjects previously treated with triheptanoin will continue to dose at approximately 35% of total daily calories (~1-4g/kg/day, depending on age).
  Schedule B: Subjects who are naïve to triheptanoin will begin a 2-week fixed titration schedule up until they have reached 35% of total daily calories (~1-4 g/kg/day depending on age). If a subject has not reached the target of 35% of total daily calories, by the end of the 2-week fixed titration period, dose titration should continue until achieved or until the maximally tolerated dose has been established.

SUMMARY:
This study is being done to assess the safety and long-term efficacy of triheptanoin in pediatric patients with Glut1 DS over a 5-year treatment period. Glut 1 is a protein that helps transport glucose to the brain. Glucose is the brain's primary source of energy. Glut 1 DS prevents this protein from being effectively produced, causing deprivation of energy to the neurons of the of the brain.

Glut1 DS is a severely debilitating disease characterized by seizures, developmental delay and movement disorder. There are currently no approved treatments specific to Glut1 DS. Treatment generally includes medications for control of seizures. The use of a ketogenic diet can be effective in controlling seizures when medications are ineffective or provide insufficient control. However, the ketogenic diet may be very difficult for patients to maintain for long periods of time, and there may be negative secondary long-term effects of ketogenic diet.. Triheptanoin is metabolized to molecules that can provide an alternative energy source to the brain, and appears to help in controlling seizures without many of the difficulties of the ketogenic diet.

Eligible patients may be those who have been diagnosed with GLUT1 DS, and have discontinued or are not currently on ketogenic diet, or are able to tolerate triheptanoin if they have been treated or are currently being treated with triheptanoin and do not qualify for any other clinical trial.

DETAILED DESCRIPTION:
Triheptanoin is proposed for the treatment of seizures in glucose transporter type-1 deficiency syndrome (Glut1 DS). Glut1 DS is a rare disease with an estimated US prevalence of ~3,300.

The proposed study is an open-label study to assess the safety and long-term efficacy of triheptanoin in patients with Glut1 DS over a 5-year treatment period. Eligible patients may be those who are able to tolerate triheptanoin if they have been treated or are currently being treated with triheptanoin and do not qualify for any other clinical trial. Subjects previously treated with triheptanoin will continue to dose at approximately 35% of total daily calories (~1-4g/kg/day, depending on age). Subjects who are naïve to triheptanoin will begin a 2-week fixed titration schedule up until they have reached 35% of total daily calories.

The primary objective of the study is to evaluate the safety of triheptanoin via adverse event rates and laboratory values. The secondary objective is to evaluate the long-term efficacy of triheptanoin as measured by the change in seizure frequency from historical baseline.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in this study must meet all of the following criteria:

1. Patients with GLUT1 DS by physician diagnosis
2. Males and females, aged 1 to 50 years
3. Allowed to be on concomitant AEDs
4. Patients are able to tolerate triheptanoin if they have been (or are currently being) treated with this medication
5. Must, in the opinion of the investigator, be willing and able to comply with study procedures and schedule
6. Provide written assent (if appropriate) and written informed consent by a Legally Authorized Representative (LAR) after the nature of the study has been explained, and prior to any research-related procedures
7. Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study
8. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study

Exclusion Criteria:

Individuals who meet any of the following exclusion criteria will not be eligible to participate in the study:

1. Patients and their Legally Authorized Representatives (as appropriate) not willing or able to give written or verbal assent or written informed consent.
2. Concomitant administration of a ketogenic diet for the treatment of GLUT1 deficiency
3. Concomitant administration of valproic acid
4. In the Investigator's opinion, the patient may not be compliant
5. Pregnant or breastfeeding an infant at screening
6. Has a concurrent disease or condition, or laboratory abnormality that, in the view of the Investigator, places the subject at high risk for adverse events, or introduces additional safety concerns
7. History of or current suicidal ideation, behavior and attempts
8. Patient qualifies for any other clinical trial designed to progressively evaluate the safety and efficacy of triheptanoin as approved by the FDA under a separate IND which is open at Cook Children's

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-20; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Lacy, MD, Principal Investigator — Cook Children's Medical Center
Locations (1):
- Cook Childrens Medical Center, Fort Worth, Texas, United States

REFERENCES:
- [Background] Johnson W Jr; Cosmetic Ingredient Review Expert Panel. Final report on the safety assessment of trilaurin, triarachidin, tribehenin, tricaprin, tricaprylin, trierucin, triheptanoin, triheptylundecanoin, triisononanoin, triisopalmitin, triisostearin, trilinolein, trimyristin, trioctanoin, triolein, tripalmitin, tripalmitolein, triricinolein, tristearin, triundecanoin, glyceryl triacetyl hydroxystearate, glyceryl triacetyl ricinoleate, and glyceryl stearate diacetate. Int J Toxicol. 2001;20 Suppl 4:61-94. PMID 11800053
- [Background] Pearson TS, Akman C, Hinton VJ, Engelstad K, De Vivo DC. Phenotypic spectrum of glucose transporter type 1 deficiency syndrome (Glut1 DS). Curr Neurol Neurosci Rep. 2013 Apr;13(4):342. doi: 10.1007/s11910-013-0342-7. PMID 23443458
- [Background] Pong AW, Geary BR, Engelstad KM, Natarajan A, Yang H, De Vivo DC. Glucose transporter type I deficiency syndrome: epilepsy phenotypes and outcomes. Epilepsia. 2012 Sep;53(9):1503-10. doi: 10.1111/j.1528-1167.2012.03592.x. Epub 2012 Jul 19. PMID 22812641
- [Background] Roe CR. Inherited disorders of mitochondrial fatty acid oxidation: a new responsibility for the neonatologist. Semin Neonatol. 2002 Feb;7(1):37-47. doi: 10.1053/siny.2002.0097. PMID 12069537
- [Background] Kinman RP, Kasumov T, Jobbins KA, Thomas KR, Adams JE, Brunengraber LN, Kutz G, Brewer WU, Roe CR, Brunengraber H. Parenteral and enteral metabolism of anaplerotic triheptanoin in normal rats. Am J Physiol Endocrinol Metab. 2006 Oct;291(4):E860-6. doi: 10.1152/ajpendo.00366.2005. Epub 2006 May 16. PMID 16705058
- [Background] Deng S, Zhang GF, Kasumov T, Roe CR, Brunengraber H. Interrelations between C4 ketogenesis, C5 ketogenesis, and anaplerosis in the perfused rat liver. J Biol Chem. 2009 Oct 9;284(41):27799-27807. doi: 10.1074/jbc.M109.048744. Epub 2009 Aug 8. PMID 19666922
- [Background] Gu L, Zhang GF, Kombu RS, Allen F, Kutz G, Brewer WU, Roe CR, Brunengraber H. Parenteral and enteral metabolism of anaplerotic triheptanoin in normal rats. II. Effects on lipolysis, glucose production, and liver acyl-CoA profile. Am J Physiol Endocrinol Metab. 2010 Feb;298(2):E362-71. doi: 10.1152/ajpendo.00384.2009. Epub 2009 Nov 10. PMID 19903863
- [Background] Marin-Valencia I, Good LB, Ma Q, Malloy CR, Pascual JM. Heptanoate as a neural fuel: energetic and neurotransmitter precursors in normal and glucose transporter I-deficient (G1D) brain. J Cereb Blood Flow Metab. 2013 Feb;33(2):175-82. doi: 10.1038/jcbfm.2012.151. Epub 2012 Oct 17. PMID 23072752
- [Background] Willis S, Stoll J, Sweetman L, Borges K. Anticonvulsant effects of a triheptanoin diet in two mouse chronic seizure models. Neurobiol Dis. 2010 Dec;40(3):565-72. doi: 10.1016/j.nbd.2010.07.017. Epub 2010 Aug 4. PMID 20691264
- [Background] Samala R, Willis S, Borges K. Anticonvulsant profile of a balanced ketogenic diet in acute mouse seizure models. Epilepsy Res. 2008 Oct;81(2-3):119-27. doi: 10.1016/j.eplepsyres.2008.05.001. Epub 2008 Jun 18. PMID 18565731
- [Background] Kim TH, Borges K, Petrou S, Reid CA. Triheptanoin reduces seizure susceptibility in a syndrome-specific mouse model of generalized epilepsy. Epilepsy Res. 2013 Jan;103(1):101-5. doi: 10.1016/j.eplepsyres.2012.09.016. Epub 2012 Nov 26. PMID 23196212
- [Background] Ataíde TdaR, de Olivera SK, da Silva FM, Vitorino Filha LGC, do N Tavares MC, Sant'Ana AEG. Toxicological analysis of the chronic consumption of diheptanoin and triheptanoin in rats. Intl J Food Sci Tech. 2009;44:484-492
- [Background] Roe CR, Sweetman L, Roe DS, David F, Brunengraber H. Treatment of cardiomyopathy and rhabdomyolysis in long-chain fat oxidation disorders using an anaplerotic odd-chain triglyceride. J Clin Invest. 2002 Jul;110(2):259-69. doi: 10.1172/JCI15311. PMID 12122118
- [Background] Roe CR, Mochel F. Anaplerotic diet therapy in inherited metabolic disease: therapeutic potential. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):332-40. doi: 10.1007/s10545-006-0290-3. PMID 16763896
- [Background] Mochel F, Duteil S, Marelli C, Jauffret C, Barles A, Holm J, Sweetman L, Benoist JF, Rabier D, Carlier PG, Durr A. Dietary anaplerotic therapy improves peripheral tissue energy metabolism in patients with Huntington's disease. Eur J Hum Genet. 2010 Sep;18(9):1057-60. doi: 10.1038/ejhg.2010.72. Epub 2010 May 26. PMID 20512158
- [Background] Baruteau J, Sachs P, Broue P, Brivet M, Abdoul H, Vianey-Saban C, Ogier de Baulny H. Clinical and biological features at diagnosis in mitochondrial fatty acid beta-oxidation defects: a French pediatric study of 187 patients. J Inherit Metab Dis. 2013 Sep;36(5):795-803. doi: 10.1007/s10545-012-9542-6. Epub 2012 Oct 3. PMID 23053472
- [Background] Goldstein A, Barone AR, DeWard SJ, Payne N, Vockley J. Triheptanoin therapy for inherited disorders of fatty acid oxidation. Mitochondrion. 2012;12(5):566
- [Background] Sparrow, SS, Cicchetti D, & Balla DA. Vineland Adaptive Behavior Scales - 2nd Edition manual. Minneapolis, MN: NCS Pearson, Inc; 2005
- [Background] Barry MJ, VanSwearingen JM, Albright AL. Reliability and responsiveness of the Barry-Albright Dystonia Scale. Dev Med Child Neurol. 1999 Jun;41(6):404-11. doi: 10.1017/s0012162299000870. PMID 10400175
- [Background] Varni JW, Burwinkle TM, Seid M. The PedsQL as a pediatric patient-reported outcome: reliability and validity of the PedsQL Measurement Model in 25,000 children. Expert Rev Pharmacoecon Outcomes Res. 2005 Dec;5(6):705-19. doi: 10.1586/14737167.5.6.705. PMID 19807613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2014 and February 2019, 20 subjects enrolled on this study. Enrollment occured in the outpatient specialty clinic offices.
Groups:
- Schedule A: Subjects previously treated with triheptanoin
  Triheptanoin: Schedule A: Subjects previously treated with triheptanoin will continue to dose at approximately 35% of total daily calories (~1-4g/kg/day, depending on age).
  Schedule B: Subjects who are naïve to triheptanoin will begin a 2-week fixed titration schedule up until they have reached 35% of total daily calories (~1-4 g/kg/day depending on age). If a subject has not reached the target of 35% of total daily calories, by the end of the 2-week fixed titration period, dose titration should continue until achieved or until the maximally tolerated dose has been established.
- Schedule B: Naïve to triheptanoin
  Triheptanoin: Schedule A: Subjects previously treated with triheptanoin will continue to dose at approximately 35% of total daily calories (~1-4g/kg/day, depending on age).
  Schedule B: Subjects who are naïve to triheptanoin will begin a 2-week fixed titration schedule up until they have reached 35% of total daily calories (~1-4 g/kg/day depending on age). If a subject has not reached the target of 35% of total daily calories, by the end of the 2-week fixed titration period, dose titration should continue until achieved or until the maximally tolerated dose has been established.
Period: Overall Study
Arm/Group | Schedule A | Schedule B
Started | 6 | 14
Completed | 6 | 8
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule A | Schedule B | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.82 (9.77) | 5.49 (3.09) | 8.29 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 14 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Seizure Count per Reporting Period [Mean (Full Range); unit: seizures] — Population: The screening visit was waived for some subjects for whom a treatment gap would have been clinically unsafe. Thus baseline seizure data were not collected prospectively for those individuals.
  seizures
    number analyzed (Participants) | 5 | 12 | 17
    (all) | 23.8 [0 to 106] | 170.7 [0 to 974] | 127.5 [0 to 974]
Barry Albright Dystonia Scale [Mean (Full Range); unit: units on a scale] — The Barry-Albright Dystonia Scale is a 5-point ordinal scale that was designed to assess dystonia in 8 body regions: eyes, mouth, neck, trunk, and the four extremities. The score in each region is rated 0 (no dystonia) to 4 (severe dystonia.) The minimum score is 0 and the maximum scale is 32 and is the sum of all of the regions measured.
  units on a scale | 8.5 [0 to 20] | 7.8 [0 to 22] | 8 [0 to 22]
PedsQL Physical Health Summary Score [Mean (Full Range); unit: units on a scale] — The PedsQL (Pediatric Quality of Life) was designed to measure perceived health-related quality of life in pediatric patients with chronic health conditions. The Generic Core scale includes assessment of physical, emotional, social, and school functioning. The summary scores are: Total Quality of Life Score, Physical Health Summary Score (avg of physical functioning), and Psychosocial Health Summary Score (avg of emotional, social, and school items). Items (5-point scale) are reversed scored and transformed to a 0-100 scale so higher scores are better. https://www.pedsql.org/about_pedsql.html
  units on a scale | 48.1 [5 to 100] | 70.8 [45 to 100] | 55.26 [5 to 100]
PedsQL Psychosocial Health Summary Score [Mean (Full Range); unit: units on a scale] — The PedsQL (Pediatric Quality of Life) was designed to measure perceived health-related quality of life in pediatric patients with chronic health conditions. The Generic Core scale includes assessment of physical, emotional, social, and school functioning. The summary scores are: Total Quality of Life Score, Physical Health Summary Score (avg of physical functioning), and Psychosocial Health Summary Score (avg of emotional, social, and school items). Items (5-point scale) are reversed scored and transformed to a 0-100 scale so higher scores are better. https://www.pedsql.org/about_pedsql.html
  units on a scale | 64.7 [42.5 to 90] | 78.6 [65 to 95] | 69.1 [42.5 to 95]

OUTCOME MEASURES:

1. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 13 Weeks
Description: A seizure diary was used to track date, type, number, and unusual presentation of seizures. Subjects were given a seizure diary at screening to record daily seizure activity for incremental periods of time. Unless otherwise waived, subjects complete this form daily during the screening period and for two weeks prior to each subsequent study visit.
Time Frame: Baseline and 13 weeks
Population: The number analyzed over time reflects both subject drop out and subjects that failed to record seizure counts during the respective reporting period.
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 5 | 12
seizures/two weeks | 4.4 [-10 to 22] | 189.5 [-228 to 2420]

2. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 26 Weeks
Description: A seizure diary was used to track date, type, number, and unusual presentation of seizures. Subjects were given a seizure diary at screening to record daily seizure activity for incremental periods of time. Unless otherwise waived, subjects complete this form daily during the screening period and for two weeks prior to each subsequent study visit. The table below represents the change in seizure frequency from baseline for each time point.
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 5 | 6
seizures/two weeks | -5.6 [-25 to 8] | -78 [-265 to 0]

3. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 1 Year
Description: as for outcome 2
Time Frame: Baseline and one yr
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 4 | 6
seizures/two weeks | -6.5 [-15 to 0] | -110.5 [-331 to 0]

4. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 18 Months
Description: as for outcome 2
Time Frame: Baseline and 18 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 5 | 6
seizures/two weeks | -5.8 [-20 to 2] | -112.7 [-340 to 3]

5. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 2 Years
Description: as for outcome 2
Time Frame: Baseline and two yrs
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 4 | 4
seizures/two weeks | -6 [-39 to 5] | -61.25 [-245 to 0]

6. Primary Outcome: Reported Change in Seizures Frequency From Baseline at 3 Years
Description: as for outcome 2
Time Frame: Baseline and three yrs
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 4 | 3
seizures/two weeks | -0.8 [-12 to 19] | -77 [-231 to 0]

7. Primary Outcome: Reported Change in Seizure Frequency From Baseline at 4 Years
Description: as for outcome 2
Time Frame: Baseline and four yrs
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 3 | 3
seizures/two weeks | -8.3 [-26 to 1] | -80.3 [-241 to 0]

8. Primary Outcome: Reported Change in Seizure Frequency From Baseline at 5 Years
Description: as for outcome 2
Time Frame: Baseline and five yrs
Population: as for outcome 1
Measure: Mean (Full Range); unit: seizures/two weeks
Arm/Group | Schedule A | Schedule B
Number analyzed (Participants) | 1 | 0
seizures/two weeks | 23 [23 to 23] |

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected for the duration of study participation for each subject from baseline through study completion or discontinuation. The longest subject participation was 5 years, 3 months.
Arm/Group | Schedule A | Schedule B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/14
Other Adverse Events (participants affected / at risk) | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule A (N=6) | Schedule B (N=14)
Prolonged generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Status Epilepticus (Nervous system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule A (N=6) | Schedule B (N=14)
Otalgia (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hirsutism (Endocrine disorders) | 1 (1) | 0 (0)
Conjuctivitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 8 (8)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 12 (14)
Emesis (Gastrointestinal disorders) | 1 (1) | 11 (19)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal Leakage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3)
Fever (General disorders) | 2 (3) | 5 (6)
Lethargy (General disorders) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 0 (0) | 1 (1)
Acute Pharyngitis (Infections and infestations) | 0 (0) | 2 (3)
Acute Tonsillitis (Infections and infestations) | 0 (0) | 1 (2)
Acute Viral Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Croup (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (5)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 5 (5)
Rhinovirus (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Stomach Virus (Infections and infestations) | 2 (2) | 1 (1)
Strep Throat (Infections and infestations) | 0 (0) | 3 (3)
Virus (Infections and infestations) | 0 (0) | 1 (1)
Fall-Witnessed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture Of Left Wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Nasal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right Arm Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right Hand Index And Middle Finger Buckle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Right Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Decreased Hematocrit (Investigations) | 1 (1) | 0 (0)
Elevated ALT (Investigations) | 0 (0) | 1 (1)
Increased Ast (Investigations) | 0 (0) | 1 (1)
Weight Gain (Investigations) | 1 (1) | 5 (5)
Weight Loss (Investigations) | 0 (0) | 1 (1)
Decrease Carbondioxide (Investigations) | 0 (0) | 1 (1)
Decreased Serum Carbon Dioxide (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 9 (11)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hand Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Balance Issues (Nervous system disorders) | 0 (0) | 1 (3)
Blurred Vision (Nervous system disorders) | 0 (0) | 1 (2)
Convulsive Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Impulsive Behavior (Nervous system disorders) | 0 (0) | 1 (1)
Increased Seizures (Nervous system disorders) | 0 (0) | 2 (2)
Lost Ability To Independently Walk (Nervous system disorders) | 0 (0) | 1 (1)
Poor Balance (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Worsening Paroxysmal Exercise Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Excessive Daytime Sleepiness (Psychiatric disorders) | 0 (0) | 1 (1)
Hyperactivity (Psychiatric disorders) | 0 (0) | 1 (1)
Hyperactivity (Adhd) (Psychiatric disorders) | 0 (0) | 1 (1)
Inattention (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Moodiness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep Difficulties (Psychiatric disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seasonal Allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Viral Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chin Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash-Right Leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scalp Laceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Scale Hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contusion of Left Foot (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT02036853/Prot_SAP_000.pdf